CLINICAL TRIAL: NCT02529540
Title: WEAR (Wearability and Evaluation of Adjustable Refraction) III: A Randomized Non-inferiority Trial of Children's Wear of Adjustable Glasses
Brief Title: WEAR (Wearability and Evaluation of Adjustable Refraction) III
Acronym: WEARIII
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sun Yat-sen University (Other)
Collaborators: Gaozhou Hospital of Traditional Chinese Medicine (Other); Xinyi traditional Chinese medicine hospital (Unknown)
Responsible Party: Principal Investigator, Congdon Nathan, Professor, MD,MPH, Sun Yat-sen University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: ZOC-WEAR 3
Record Dates: First submitted 2015-08-16; First posted 2015-08-20 (Estimated); Last update posted 2018-10-15 (Actual); Status verified 2018-10

CONDITIONS: Myopia
Keywords: Myopia; self-refraction; glasses; spectacles
MeSH Terms: conditions — Myopia

STUDY DESIGN:
Intervention Model Description: This is a randomized non-inferiority trial, and the margin of the non-inferiority is 20%.
Oversight: Data Monitoring Committee: No

ARMS (3):
- Group 1 (Other): Self-refraction with adjustable glasses
  Interventions: Other: Adjustable glasses
- Group 2 (Other): Subjective refraction by an expert refractionist after auto refraction and receiving custom standard glasses
  Interventions: Other: Custom standard glasses
- Group 3 (Other): Subjective refraction by an expert refractionist after auto refraction and receiving ready-made glasses
  Interventions: Other: Ready-made glasses

INTERVENTIONS:
Other: Adjustable glasses — The glasses will be used for refraction and wearing within professional instructions.
  Arms: Group 1
Other: Custom standard glasses — The custom standard glasses are made by the traditional standards after refraction.
  Arms: Group 2
Other: Ready-made glasses — The glasses have been made already before the refraction in the hospital. And they will be chosen by prescription after refraction.
  Arms: Group 3

SUMMARY:
Two-month randomized trial comparing three groups.

DETAILED DESCRIPTION:
Two-month randomized non-inferiority trial (the margin of non-inferiority is 20%) comparing three groups: self-refraction with adjustable glasses, receiving adjustable glasses; subjective refraction by an expert refractionist after computer optometry and receiving custom standard glasses; subjective refraction by an expert refractionist after computer optometry and receiving ready-made glasses. The main outcome of this study is the rate of glasses wear on twice-weekly covert evaluation by head teachers. And the continuous teacher assessment of wearing study glasses will be calculated as the number of times wearing glasses/ Total number of separate observations.

ELIGIBILITY:
Inclusion Criteria:

* 11-16 years old middle school students from two locations in Guangdong Province.
* With ≤ -1.00 Diopter of myopic refractive error in each eye.
* With uncorrected vision ≤ 6/12 in both eyes thought to be due to refractive error (that is, correctable to at least 6/7.5 with subjective refraction by an optometrist).
* With informed consents(There are two types of informed consents. One of them is whether the parents of the students agree their kids to participate in the project. The other informed consent is whether the parents agree their kids to have the cycloplegic refraction. If the students were admitted to participate in project but without being agreed to have cycloplegic refraction by their parents , they would have non cycloplegic retinoscopy.).

Exclusion Criteria:

* Those corrected VA can not up to 6/7.5 with subjective refraction by an optometrist.
* Those with significant strabismus or vision abnormality (keratopathy, cataract, vitreous macular diseases ), or with vision deficiency ( amblyopia ) children are to be excluded.
* Children developing acquired vision problems other than myopia.

Ages: 11 Years to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 324 (Actual)
Dates: Start 2015-09-01 (Actual); Primary Completion 2016-06-01 (Actual); Study Completion 2016-06-01 (Actual)

PRIMARY OUTCOMES:
Wearing spectacles proportion | 5 months after the start of the project
  The participators in each group may have the different wearing spectacles proportion.

SECONDARY OUTCOMES:
The quality of life after wearing glasses(questionnaires) | 5 months after the start of the project
  The quality of life will be learned by questionnaires

OTHER OUTCOMES:
Evaluation of the user's subjective impression（questionnaires） | 5 months after the start of the project
  Evaluation of the user's subjective impression for the three type of glasses will be learned by questionnaires.
Damaged condition of the glasses | 5 months after the start of the project
  The glasses may be damaged during use. At the end of project, every user will have have a questionnaire about damaged condition of glasses, such as missing screws, having scratches on the surface of lens and so on.

CONTACTS AND LOCATIONS:
Overall Officials: Nathan Congdon, MD, MPH, Principal Investigator — The Key Laboratory, Zhongshan Ophthalmic Center, Sun Yat-sen University

REFERENCES:
- [Background] He M, Zeng J, Liu Y, Xu J, Pokharel GP, Ellwein LB. Refractive error and visual impairment in urban children in southern china. Invest Ophthalmol Vis Sci. 2004 Mar;45(3):793-9. doi: 10.1167/iovs.03-1051. PMID 14985292
- [Background] He M, Zheng Y, Xiang F. Prevalence of myopia in urban and rural children in mainland China. Optom Vis Sci. 2009 Jan;86(1):40-4. doi: 10.1097/OPX.0b013e3181940719. PMID 19104465
- [Background] Li L, Lam J, Lu Y, Ye Y, Lam DS, Gao Y, Sharma A, Zhang M, Griffiths S, Congdon N. Attitudes of students, parents, and teachers toward glasses use in rural China. Arch Ophthalmol. 2010 Jun;128(6):759-65. doi: 10.1001/archophthalmol.2010.73. PMID 20547954
- [Background] He M, Congdon N, MacKenzie G, Zeng Y, Silver JD, Ellwein L. The child self-refraction study results from urban Chinese children in Guangzhou. Ophthalmology. 2011 Jun;118(6):1162-9. doi: 10.1016/j.ophtha.2010.10.003. Epub 2011 Jan 12. PMID 21232802
- [Background] Zhou Z, Zeng J, Ma X, Pang X, Yi H, Chen Q, Meltzer ME, He M, Rozelle S, Congdon N. Accuracy of rural refractionists in western China. Invest Ophthalmol Vis Sci. 2014 Jan 7;55(1):154-61. doi: 10.1167/iovs.13-13250. PMID 24327616
- [Derived] Wang CY, Zhang G, Tang B, Jin L, Huang W, Wang X, Chen T, Zhu W, Xiao B, Wang J, Zhou Z, Tang Z, Liang Y, Crescioni M, Wilson D, McAneney H, Silver JD, Moore B, Congdon N. A Randomized Noninferiority Trial of Wearing Adjustable Glasses versus Standard and Ready-made Spectacles among Chinese Schoolchildren: Wearability and Evaluation of Adjustable Refraction III. Ophthalmology. 2020 Jan;127(1):27-37. doi: 10.1016/j.ophtha.2019.08.002. Epub 2019 Aug 14. PMID 31543351